CLINICAL TRIAL: NCT02308982
Title: A Phase III Multi-centre Randomised, Double Blind, Placebo Controlled Trial to Assess the Role of Intravenous Immunoglobulin in the Management of Children With Encephalitis
Brief Title: Investigating the Role of Early Intravenous Immunoglobulin Treatment for Children With Encephalitis
Acronym: IgNiTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); CSL Behring (Industry); University of Liverpool (Other); University College London Hospitals (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OVG 2014/05
Record Dates: First submitted 2014-12-01; First posted 2014-12-05 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2022-09

CONDITIONS: Encephalitis
Keywords: encephalitis; meningoencephalitis; encephalomyelitis; brain inflammation; intravenous immunoglobulin; randomised controlled trial; Central Nervous System Diseases; Central Nervous System Infection
MeSH Terms: conditions — Encephalitis; Meningoencephalitis; Encephalomyelitis; Central Nervous System Diseases; Central Nervous System Infections | interventions — Immunoglobulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous immunoglobulin (Active Comparator): Intravenous immunoglobulin: 1g/kg per day for 2 consecutive days
  Interventions: Drug: Immunoglobulins, Intravenous (Privigen)
- Placebo (Placebo Comparator): Equivalent volume to 1g/kg of IVIG per day for 2 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Immunoglobulins, Intravenous (Privigen)
  Other Names: Privigen
  Arms: Intravenous immunoglobulin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a phase III multi-centre randomised, double blind, placebo controlled trial to assess the role of intravenous immunoglobulin in the treatment of children with encephalitis. The primary objective is to find out whether early use of IVIG treatment improves neurological outcomes of children with encephalitis.

308 children with encephalitis, aged 6 weeks to 16 years will be recruited in 30 hospitals in the United Kingdom. Participants will be randomised to receive two doses of IVIG or matching placebo in addition to other standard treatments, within the first five days of hospital admission.

Each participant will be followed up for 12 months. During this period, information on clinical, radiological and laboratory investigations will be collected. Neurological outcomes will be assessed by the use of questionnaires at 6 and 12 months, and a neuropsychological assessment at 12 months.

DETAILED DESCRIPTION:
Encephalitis is a syndrome of neurological dysfunction caused by inflammation of the brain parenchyma, resulting in altered mental status, seizures, and/or focal neurologic deficits, usually accompanied by laboratory and radiological evidence of brain inflammation. The worldwide annual incidence of encephalitis ranges from 3.5 to 7.4 per 100,000, rising to 16 per 100,000 in children. In the United Kingdom, Public Health England (formerly the Health Protection Agency) reports an annual rate of 1.5 cases per 100,000 in the general population and 2.8 per 100,000 in children, with the highest incidence in infants under 1 year of age of 8.7 per 100,000.

Despite the use of current standard treatments, mortality of 7-10% and morbidity of up to 50% are still being reported. Encephalitis also imposes a substantial economic and resource burden on healthcare services. Strategies to reduce the disability in patients with encephalitis are therefore required.

There is increasing evidence from case reports of a beneficial role of IVIG treatment in encephalitis. However, in clinical practice, the use of IVIG in encephalitis varies. The variation in practice is in most part due to a lack of class 1 evidence to support the use of IVIG in encephalitis. For the immune mediated forms of encephalitis, IVIG is typically used after inevitable delay (by weeks in some cases) while alternative diagnoses are being excluded, or a definitive diagnosis is obtained. In other cases, IVIG is used usually as a last treatment option where clinical improvement is slow. Again, this is usually after several days from hospital admission. Delays in the institution of appropriate treatment in encephalitis may contribute to the high rate of morbidity and mortality, prolonged hospitalisation and associated costs from encephalitis. In particular, it is currently unknown whether wider use of IVIG in infectious encephalitis and earlier use in immune-mediated encephalitis could alter the outcome of this group of conditions.

This study will fill in the evidence gap on the potential benefit of IVIG in reducing disease burden in children with encephalitis. The trial also aims to generate evidence to inform clinical decision making in the National Health Service (NHS) and provide added value to the NHS by addressing healthcare, quality of life and productivity costs of this expensive and resource limited product.

ELIGIBILITY:
Inclusion Criteria:

1. 6 weeks to 16 years of age (day before 17th birthday) AND
2. Acute (within 24 hours) or sub-acute (between 24 hours and 4 weeks) onset of altered mental state (reduced or altered conscious level, irritability, altered personality or behaviour, lethargy) not attributable to a metabolic cause AND
3. At least two of:

   1. fever > 38 degrees Celsius within 72 hours before or after presentation to hospital
   2. brain imaging evidence consistent with encephalitis or immune-mediated encephalopathy that is either new from prior studies or appears acute in onset
   3. CSF pleocytosis > 4 white blood cells per microlitre
   4. generalised or partial seizures not fully attributable to a pre-existing seizure disorder
   5. new onset focal neurological signs (including movement disorders) for > 6 hours
   6. abnormality on EEG that is consistent with encephalitis and not clearly attributable to another cause AND
4. Parent/guardian/legal representative able to give informed consent

Exclusion Criteria:

* high clinical suspicion of bacterial meningitis or TB meningitis (for example: presence of frankly purulent CSF; CSF WBCs >1000/microlitre; bacteria on Gram stain and/or culture)
* Traumatic brain injury
* Known metabolic encephalopathy
* toxic encephalopathy (i.e. encephalopathy secondary to exposure to intoxicants, including alcohol, prescription or recreational drugs)
* hypertensive encephalopathy/posterior reversible encephalopathy syndrome
* pre-existing demyelinating disorder; pre-existing antibody mediated CNS disorder; pre-existing CSF diversion
* ischaemic or haemorrhagic stroke
* children with a contra-indication to IVIG or albumin (i.e. history of anaphylactic reaction to IVIG or albumin, known IgA deficiency and history of hypersensitisation)
* Known hypercoagulable state
* significant renal impairment defined as GFR of 29mls/min/1.73m2 and below (Chronic Kidney Disease Stage 4)
* Known hyperprolinaemia
* Known to be pregnant
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
* participants who are being actively followed up in another research trial involving an investigational medicinal product
* Administration of study drug not feasible within 120 hours from hospital admission as determined by the study team
* Any other condition which, in the opinion of the investigator, may interfere with the ability to fulfil study requirements, especially relating to the primary objective of the study (this includes plans to be outside the UK for more than 12 months after enrolment)

Ages: 6 Weeks to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2016-01; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Good recovery", defined by GOS-E-Peds score 2 or lower at 12 months post randomisation | Up to 12 Months after randomization
  Compare neurological outcomes between children with encephalitis who have been treated with IVIG and those who have received matching placebo

SECONDARY OUTCOMES:
Brain MRI scan changes | Up to 6 months after randomization
  assessment of using lesion resolution presence of new lesions distribution of persisting disease
Local and systemic adverse events of interest and serious adverse events | Up to 6 months after randomization
  Collection of all serious and non-serious adverse events, including full blood count check 24-48 hours after the second dose of the study drug to monitor for possible haemolysis with IVIG treatment.
Clinical outcomes such as length of hospitalisation, need for intensive care admission, duration of invasive ventilation, frequency of seizures and need for anti-epileptic treatment | Up to 12 months after randomization
  Review neurological examination findings as documented in clinical records, identify the need for, and duration of ventilation (for ventilated participants). Also review results of laboratory tests and brain MRI scans which would possibly elongate hospitalisation.
Presence of auto-antibodies in blood and/or cerebrospinal fluid (CSF) | Up to 12 Months after randomization
  Obtain scavenged blood and CSF during the entire study period: prior to and after enrolment; for auto-antibody evaluation.

OTHER OUTCOMES:
To explore clinically relevant neuroimaging predictors | Up to 12 Months after randomization
  Correlate MRI findings with the primary and secondary outcomes
To explore predictors of neurological outcomes in children with encephalitis | Up to 12 Months after randomization
  Correlate clinical and laboratory parameters with neurological outcomes
To explore radiological patterns associated with different types of encephalitis | Up to 12 Months after randomization
  Further analysis that will include using a systematic structured study proforma designed to capture data that would then subsequently be used to aid in:
  (i) identifying imaging subtypes of different encephalitides for example infectious vs. demyelinating vs. autoimmune
  (ii) identifying clinically relevant neuroimaging predictors.
To understand the host inflammatory pathways in encephalitis | Up to 12 Months after randomization
  (i) Analysis of gene expression in whole blood before and after study treatment
  (ii) Identification of specific DNA sequence and structural genetic variants in patients with encephalitis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Pollard, FRCPCH, PhD, Principal Investigator — University of Oxford
Locations (25):
- United Kingdom (25):
  - Grampian Health Board, Aberdeen
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Heart of England NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Tayside Health Board, Dundee
  - Lothian Health Board, Edinburgh
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Guy's and St Thomas's NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Great Ormond Street Hospital, London
  - Barts Health NHS Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - The Pennine Acute Hospitals NHS Trust, Manchester
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Sheffield Children's NHS Foundation Trust, Sheffield
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent
  - Royal Cornwall Hospitals NHS Trust, Truro
  - York Teaching Hospital NHS Foundation Trust, York

REFERENCES:
- [Background] Iro MA, Sadarangani M, Absoud M, Chong WK, Clark CA, Easton A, Gray V, Kneen R, Lim M, Pike M, Solomon T, Vincent A, Willis L, Yu LM, Pollard AJ. ImmunoglobuliN in the Treatment of Encephalitis (IgNiTE): protocol for a multicentre randomised controlled trial. BMJ Open. 2016 Nov 3;6(11):e012356. doi: 10.1136/bmjopen-2016-012356. PMID 27810972
- [Derived] Hill M, Iro M, Sadarangani M, Absoud M, Cantrell L, Chong K, Clark C, Easton A, Gray V, Kneen R, Lim M, Liu X, Pike M, Solomon T, Vincent A, Willis L, Yu LM, Pollard AJ; IgNiTE study team. Intravenous immunoglobulin treatment in childhood encephalitis (IgNiTE): a randomised controlled trial. BMJ Open. 2023 Nov 9;13(11):e072134. doi: 10.1136/bmjopen-2023-072134. PMID 37945292
- See also: Intravenous immunoglobulin treatment in childhood encephalitis (IgNiTE): a randomised controlled trial — https://bmjopen.bmj.com/content/13/11/e072134.long
- See also: ImmunoglobuliN in the Treatment of Encephalitis (IgNiTE): protocol for a multicentre randomised controlled trial — https://pubmed.ncbi.nlm.nih.gov/27810972/